CLINICAL TRIAL: NCT00891865
Title: Viral Triggers of Alloimmunity and Autoimmunity in Pediatric Lung Transplantation (CTOTC-03)
Brief Title: Viral Triggers in Pediatric Lung Transplantation
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOTC-03
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Lung Transplant; Bronchiolitis Obliterans; Obliterative Bronchiolitis
Keywords: lung transplant; BOS; OB; Respiratory Viral Infection (RVI); Lung disease
MeSH Terms: conditions — Bronchiolitis Obliterans; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and nasopharyngeal samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pediatric lung transplantation

SUMMARY:
The purpose of this study is to determine whether respiratory viral infections increase the risk of bronchiolitis obliterans syndrome (BOS), obliterative bronchiolitis (OB), death, or retransplantation in children who have received lung transplants.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian willing and able to provide informed consent
* Participant of first single or bilateral heart-lung transplant

Exclusion Criteria:

* Recipient of multi-organ transplant (aside from heart-lung)
* Condition or characteristic which in the opinion of the investigator makes the participant unlikely to complete the study

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients undergoing lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2009-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The earliest time to BOS or OB, retransplantation or death | Within 24 months of transplant

SECONDARY OUTCOMES:
Time to each of the following events: BOS or OB, retransplantation or death | Within 24 months of transplant

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Sweet, MD, PhD, Principal Investigator — Washington University School of Medicine; Lara Danziger-Isakov, MD, MPH, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (6):
- United States (6):
  - Stanford University, Palo Alto, California
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Background] Hayes D Jr, Ballard HO. Saber-sheath trachea in a patient with bronchiolitis obliterans syndrome after lung transplantation. Chron Respir Dis. 2009;6(1):49-52. doi: 10.1177/1479972308099990. PMID 19176714
- [Background] Sweet SC. Pediatric lung transplantation. Proc Am Thorac Soc. 2009 Jan 15;6(1):122-7. doi: 10.1513/pats.200808-095GO. PMID 19131537
- [Background] Vos R, Vanaudenaerde BM, De Vleeschauwer SI, Van Raemdonck DE, Dupont LJ, Verbeken EK, De Wever W, Verleden GM. Follicular bronchiolitis: a rare cause of bronchiolitis obliterans syndrome after lung transplantation: a case report. Am J Transplant. 2009 Mar;9(3):644-50. doi: 10.1111/j.1600-6143.2008.02518.x. Epub 2009 Feb 3. PMID 19191770
- [Background] Yun JJ, Mason DP. Lung transplantation: past, present, and future. Minerva Chir. 2009 Feb;64(1):37-44. PMID 19202534
- [Result] Sweet SC, Chin H, Conrad C, Hayes D Jr, Heeger PS, Faro A, Goldfarb S, Melicoff-Portillo E, Mohanakumar T, Odim J, Schecter M, Storch GA, Visner G, Williams NM, Kesler K, Danziger-Isakov L. Absence of evidence that respiratory viral infections influence pediatric lung transplantation outcomes: Results of the CTOTC-03 study. Am J Transplant. 2019 Dec;19(12):3284-3298. doi: 10.1111/ajt.15505. Epub 2019 Jul 25. PMID 31216376